CLINICAL TRIAL: NCT03019458
Title: MINGO Supplemental Trial in X-linked Dystonia Parkinsonism Patients: A Prospective Randomized, Open-labeled, Parallel Group Trial
Brief Title: MINGO Supplemental Trial in X-linked Dystonia-Parkinsonism Patients
Acronym: MINGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunshine Care Foundation (Other)
Collaborators: Jose R. Reyes Memorial Medical Center (Other Government); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MINGO-001
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: X-Linked Dystonia Parkinsonism
Keywords: prospective randomized trial
MeSH Terms: conditions — Dystonia 3, Torsion, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINGO (Experimental): MINGO is a supplement consisting of local ingredients such as moringa, rice and mung beans, which can be added to any type of edible paste, food, and liquid. The experimental group is required to take 6 sachets per day for 12 weeks in addition to their regular diet. They are required to keep a daily food diary
  Interventions: Dietary Supplement: MINGO
- Control (No Intervention): The control group is required to eat their normal diet. They are also required to keep a daily food diary.

INTERVENTIONS:
Dietary Supplement: MINGO — 6 20oz sachets will be taken daily by intervention group
  Arms: MINGO

SUMMARY:
To see whether MINGO, a food supplement, will be able to lessen the drastic weight loss seen among X-linked Dystonia Parkinsonism patients.

DETAILED DESCRIPTION:
X-linked dystonia parkinsonism (XDP, formerly known as DYT3) occurs primarily in Filipino males and is characterized by neurodegenerative dystonia and parkinsonism. It is currently recognized to have wide phenotypic variability relating to age of onset, location of disease onset and rate of severity/disease progression. Most patients begin with focal dystonia that generalizes with the development of parkinsonism later in disease course. XDP patients suffer from severe nutritional loss due to symptoms such as dysphagia, loss of appetite, and consistently high metabolic requirements brought about by their movement disorder. Approximately 79% of patients with XDP have experienced rapid weight loss since the onset of their disease. It is the aim of the researchers to assess the clinical usefulness of adding a nutritional supplement to the daily dietary needs of these patients.

MINGO is a supplement consisting of local ingredients such as moringa, rice and mung beans, which can be added to any type of edible paste, food, and liquid. Mingo has gained popularity as an emergency food in disaster relief operations due to the ease of its preparation, its high nutritional value and relatively low price. For the last two years, it has also been used as an agent for nutritional build up in malnourished populations of children. This study will provide valuable information on whether patients with XDP can increase their weight by consuming MINGO, which will lead to improvements in the patients' medical care and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Subject is above the age of 18
* Positive Diagnosis of XDP by movement disorder specialist/fellow
* Subject with a yes response to a "supportive home environment" in the patient's most recent "doctors monthly report"
* Subject are easily accessible to passable roads and pubic transportation

Exclusion Criteria:

* Subjects who have extreme movements that prevent staff from performing BMI or MUAC measurements
* Subjects who have abnormal metabolic labs prior to the start of the study
* Subjects who are taking pharmacological or medicinal supplements that may effect weight
* Subjects who have been hospitalized within the last 2 weeks from the start of the trial
* Subjects who have a Nasogastric tube or G-tube
* Subjects with a history of other diseases that my effect weight (eg: hypo/hyperthyroidism)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Criscely L Go, MD,FPNA,DPBP, Principal Investigator — Jose R. Reyes Memorial Medical Center
Locations (1):
- Health Centrum, Roxas City, Capiz, Philippines

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MINGO: MINGO is a supplement consisting of local ingredients such as moringa, rice and mung beans, which can be added to any type of edible paste, food, and liquid. The experimental group is required to take 6 sachets per day for 12 weeks in addition to their regular diet. They are required to keep a daily food diary
  MINGO: 6 20oz sachets will be taken daily by intervention group.
  There were 24 subjects who were part of the MINGO arm.
- Control: The control group is required to eat their normal diet. They are also required to keep a daily food diary. There were a total of 26 subjects who were enrolled in the Control group
Period: Overall Study
Arm/Group | MINGO | Control
Started | 24 | 26
Completed | 24 | 25
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MINGO | Control | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (1.6) | 56.4 (1.6) | 55.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 26 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 26 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Philippines | 24 | 26 | 50
Duration of Illness [Mean (Standard Deviation); unit: years] | 9.4 (1.1) | 8.2 (1.1) | 8.8 (0.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 18.9 (0.6) | 18.2 (0.4) | 18.5 (0.4)
Mean Upper Arm Circumference (MUAC) [Mean (Standard Deviation); unit: cm] | 26.5 (0.5) | 26.5 (0.6) | 26.5 (0.4)
Burkes-Fahn-Marsden (BFM) [Mean (Standard Deviation); unit: units on a scale] — This is a scale that is done to score dystonia severity from 0 to 120 with higher numbers indicating worse outcome. A movement disorder specialist was the one who performed the scale.
  units on a scale | 44.1 (5.3) | 40.2 (4.8) | 42.1 (3.5)
Eating Assessment Tool (EAT-10) [Mean (Standard Deviation); unit: units on a scale] — EAT-10 is a subjective swallowing screening tool for dysphagia that ranges from 0-40 with higher scores meaning more difficulty in swallowing
  units on a scale | 20.0 (2.3) | 19.9 (2.6) | 19.9 (1.7)
MGH-Swallowing Screening Tool (MGH-SST) [Mean (Standard Deviation); unit: units on a scale] — MGH SST is an objective swallowing screening tool to determine the risk of aspiration from 0-5 with 5 being the highest risk to aspiration
  units on a scale | 3.8 (0.3) | 3.8 (0.3) | 3.8 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: The Body Mass Index (BMI in kg/m^2) Using a Bathroom Weighing Scale.
Description: The investigators will first take a baseline Body Mass Index in kg/m^2 for both control and intervention group, then subsequent measures every two weeks for 3 month duration of he trial. The goal of the investigators is to compare the net change in Body Mass Index in a 3 month period.
Time Frame: after baseline Body Mass Index, we will measure Body Mass Index every 2 weeks for 3 months
Population: We proposed an intention to treat analysis, so regardless of whether an XDP subject took the prescribed # of MINGO packets or not we analyzed everyone who entered the trial
Measure: Mean (95% Confidence Interval); unit: Kg/m^2
Arm/Group | MINGO | Control
Number analyzed (Participants) | 24 | 26
Kg/m^2
  baseline | 18.86 [17.66 to 20.06] | 18.17 [17.24 to 19.09]
  week 2 | 19.00 [17.75 to 20.24] | 18.31 [17.30 to 19.31]
  week 4 | 19.14 [17.91 to 20.37] | 18.27 [17.25 to 19.29]
  week 6 | 19.11 [17.90 to 20.33] | 18.06 [17.01 to 19.11]
  week 8 | 19.15 [17.89 to 20.40] | 18.24 [17.24 to 19.24]
  week 10 | 19.03 [17.77 to 20.28] | 18.05 [17.01 to 19.10]
  week 12 | 19.07 [17.83 to 20.31] | 17.95 [16.90 to 18.99]
Statistical Analysis 1: Comparison: MINGO vs Control; Test type: Superiority; p = 0.084, Mixed Models Analysis — The p value was not adjusted for multiple comparisons but rather it is the priori threshold for statistical significance at p<0.05; We adjusted for baseline Eating Assessment Tool-10 (EAT-10), MGH-Swallowing Screening Test (MGH-SST), and the Burkes-Fahn-Marsden Dysonia Scale (BFM)

2. Secondary Outcome: All Cause Mortality
Description: number of deaths in both arms at the end of the study
Time Frame: 3 months (study close out)
Population: Everyone who enrolled were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | MINGO | Control
Number analyzed (Participants) | 24 | 26
Participants | 0 | 1

3. Secondary Outcome: Number of Hospitalizations Secondary to Infectious Causes
Description: number of hospitalizations secondary to infections in both arms at the end of the study
Time Frame: 3 months (study close out)
Population: all participants were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | MINGO | Control
Number analyzed (Participants) | 24 | 26
Participants | 0 | 0

4. Secondary Outcome: Mid Upper Arm Circumference (MUAC) in cm Using a Tailor's Tape Measure
Description: It has been reported that the Mid Upper Arm Circumference is a good predictor for BMI. It will serve as an indirect measurement to the subjects' BMI
Time Frame: After baseline measurements, the investigators will measure the MUAC evey month for 3 months
Population: All participants in the trial
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | MINGO | Control
Number analyzed (Participants) | 24 | 26
cm
  baseline | 26.54 [25.39 to 27.59] | 26.54 [25.24 to 27.84]
  month 1 | 26.93 [25.86 to 28.00] | 26.58 [25.23 to 27.93]
  month 2 | 26.96 [25.85 to 28.07] | 26.69 [25.13 to 28.07]
  month 3 | 26.69 [25.41 to 27.97] | 26.62 [25.03 to 28.18]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | MINGO | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 4/24 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MINGO (N=24) | Control (N=26)
Intolerance to taking MINGO (Gastrointestinal disorders) | 4 (4) | 0 (0) — Any intolerance to taking MINGO that caused the subject to stop taking the supplement including 1 due to vomiting, 1 due to the subjective sensation to fullness, and 2 due to the fact they did not like the taste of MINGO.
GI symptoms (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A major limitation to this trial is that it was a community-based clinical trial that relied on 14 CHWs to measure the weight and MUAC due to the far distance and difficult terrain. The accuracy of subject's food diary is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT03019458/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT03019458/SAP_001.pdf